CLINICAL TRIAL: NCT02140567
Title: Syncope Prediction Study
Acronym: SPS
Status: Completed | Type: Observational
Sponsor: Medtronic BRC (Industry)
Responsible Party: Sponsor
Other Study IDs: Syncope Prediction Study; SPS (Other: sponsor)
Record Dates: First submitted 2014-04-30; First posted 2014-05-16 (Estimated); Results first posted 2018-08-27 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-02

CONDITIONS: Vasovagal Syncope
MeSH Terms: conditions — Syncope, Vasovagal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Syncope Prediction: All enrolled patients that performed the tilt table test

SUMMARY:
The purpose of this study is to perform a prospective evaluation of the vasovagal syncope prediction algorithm, called Tilt Test Analyzer, during head up tilt testing tests in one center in the United Kingdom.

DETAILED DESCRIPTION:
Vasovagal syncope (VVS) is a form of neurally-mediated reflex syncope, which is marked by a sudden fall in blood pressure with an associated fall in heart rate often resulting in syncope, head-up tilt (HUT) testing is commonly used to bring information about VVS using ECG and blood pressure monitoring with medical observation.

We developed an algorithm, called Tilt Test Analyzer, to predict VVS during HUT based on the simultaneous analysis of heart rate (RR interval), systolic blood pressure (SBP) and an indicator of autonomic modulation represented by heart rate and blood pressure variability (HRV and BPV).

The primary objective of this study is to evaluate the VVS prediction algorithm in a prospective cohort of patients in the tilt laboratory The primary endpoint is the VVS prediction algorithm performance by means of measuring the sensitivity and specificity values.

The study is designed to test if the prospective analysis of tilt-test patients can reproduce the results previously obtained in the published retrospective analysis on 1155 patients with a similar clinically relevant sensitivity and specificity.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to the center with vasovagal syncope for tilt testing.
* The patient is willing and able to cooperate with the study procedures.
* The subject or legal guardian is able to provide written informed consent

Exclusion Criteria:

* Patients under 18 years or over 90 years old.
* Women who are currently pregnant or have a positive pregnancy test.
* Patients who had a prior tilt test.
* Patients enrolled in another device or drug study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Vasovagal syncope patients
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2014-11; Primary Completion 2016-10 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: P Boon Lim, MD, Principal Investigator — Hammersmith Hospital, Imperial College Healthcare NHS Trust
Locations (1):
- Hammersmith Hospital, Imperial College Healthcare NHS Trust, London, United Kingdom

REFERENCES:
- [Derived] Virag N, Erickson M, Taraborrelli P, Vetter R, Lim PB, Sutton R. Predicting vasovagal syncope from heart rate and blood pressure: A prospective study in 140 subjects. Heart Rhythm. 2018 Sep;15(9):1404-1410. doi: 10.1016/j.hrthm.2018.04.032. Epub 2018 Apr 30. PMID 29715516

RESULTS

PARTICIPANT FLOW:
Groups:
- Syncope Prediction Study: All enrolled participants who performed a tilt test.
Period: Overall Study
Arm/Group | Syncope Prediction Study
Started | 140
Completed | 134
Not Completed | 6
Not completed — Problems with recording equipment | 6

BASELINE CHARACTERISTICS:
Population: Participants included in efficacy analysis
Groups:
- Syncope Prediction: Enrolled participants who performed tilt test and were included in efficacy analysis
Arm/Group | Syncope Prediction
Number analyzed (Participants) | 134
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.2 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92
  Male | 42

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity of the Syncope Prediction Algorithm
Description: Number of tilt-positive participants predicted in the right way by the syncope prediction algorithm
Time Frame: Tilt Test with average duration of 1 hour
Population: Number of participants with positive tilt-test
Measure: Count of Participants; unit: Participants
Groups:
- Syncope Prediction (Sensitivity): Tilt-positive participants included in the efficacy analysis
Arm/Group | Syncope Prediction (Sensitivity)
Number analyzed (Participants) | 83
Participants
  True positive | 81
  False negative | 2

2. Primary Outcome: Specificity of the Syncope Prediction Algorithm
Description: Number of tilt-negative participants identified as negative by the syncope prediction algorithm
Time Frame: Tilt Test with average duration of 1 hour
Population: Number of participants with negative tilt-test
Measure: Count of Participants; unit: Participants
Groups:
- Syncope Prediction (Specificity): Tilt-negative participants included in the efficacy analysis
Arm/Group | Syncope Prediction (Specificity)
Number analyzed (Participants) | 51
Participants
  True negative | 45
  False positive | 6

ADVERSE EVENTS:
Time Frame: 1 hour
Groups:
- Syncope Prediction: Enrolled participants who performed the tilt test
Arm/Group | Syncope Prediction
All-Cause Mortality (participants affected / at risk) | 0/140
Serious Adverse Events (participants affected / at risk) | 0/140
Other Adverse Events (participants affected / at risk) | 0/140

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No